CLINICAL TRIAL: NCT01286259
Title: Short-term Disulfiram Administration to Accelerate the Decay of the HIV Reservoir in Antiretroviral-treated HIV Infected Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 10-02648
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: HIV-1 Infection
Keywords: HIV; HAART suppressed; Disulfiram; Antabuse; Latent reservoir; Eradication; Cure
MeSH Terms: interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Open label 500mg disulfiram per day by mouth for 14 days
  Other Names: Antabuse

SUMMARY:
The purpose of this study is to determine whether a two-week course of disulfiram will reduce the HIV-1 latent reservoir in patients on highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
This study is using a new approach to try and force HIV out of its protected cellular reservoirs.

Although current therapies are effective at "killing" new viruses that are produced, they are unable to access the virus in cells which were infected before antiretroviral therapy began. HIV can remain "hidden" in a latent (or resting) form in these cells for many years. Since these infected cells can live for many years, they are thought to be the most important barrier to HIV eradication (or "cure").

Many experts believe that one way to attack latent or "hidden" HIV is to use a drug than can "turn on" the virus and hence force HIV-1 out of resting T cells. In a recent study done in the laboratory, disulfiram proved to be among the most effective drugs currently available that can reactivate latent HIV-1,

Our primary hypothesis is that disulfiram will reduce the latent reservoir of HIV-1 in patients on highly active antiretroviral therapy (HAART). Theoretically, disulfiram will force HIV to replicate (grow) and thus result in the death of the infected cell. Standard antiretroviral drugs should prevent new cells from becoming infected. The end result of this process is that the total amount of HIV in the body will decline over time.

ELIGIBILITY:
Inclusion Criteria:

* Documented continuous HAART for at least 18 months prior to study entry and on a stable regimen for at least 3 months prior to entry.
* Documented undetectable HIV viral loads for at least one year. Intermittent isolated episodes of detectable low-level viremia "blips" (> 50 but < 500 copies RNA/mL) remain eligible.
* Screening plasma HIV-1 RNA levels < 40 copies RNA/mL.
* CD4 T-cell count above 200 cells/uL for 24 weeks prior to screen.
* >90% adherence to therapy within the preceding 30 days.
* Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
* Willing to abstain from any alcohol during the two week period in which disulfiram will be administered and during the two week period immediately after disulfiram administration.

Exclusion Criteria:

* Current alcohol use disorder or hazardous alcohol use as determined by clinical evaluation.
* Current use of any drug formulation that contains alcohol or that might contain alcohol.
* Current use of tipranavir.
* Current use of maraviroc.
* Current use of warfarin.
* Intending to modify antiretroviral therapy in the next 27 weeks for any reason.
* Serious illness requiring hospitalization or parental antibiotics within preceding 3 months.
* Severe myocardial disease or coronary artery disease.
* History of psychosis.
* Clinically active hepatitis determined by the study physician; ALT or AST >3 x the upper limit of normal.
* Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drug in past 16 weeks.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Deeks, M.D., Principal Investigator — University of California, San Francisco; Adriana Andrade, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 47.5 [24 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Impact of Two Weeks of Disulfiram, as Measured by the Fold Change in the Infectious Units Per Million Cells (IUPM) Between Baseline and Week 12
Description: The size of the latent reservoir from each participant was measured by limiting dilution co-culture assay and reported as "infectious units per million cells" (IUPM).This assay measures the frequency of peripheral blood cells from which replication-competent HIV can be grown. The assay was performed at a baseline visit (two weeks before dosing began) and week 12 (10 weeks after the last dose). The primary outcome was the fold-change in IUPM before and after disufiram.
Time Frame: 12 weeks
Population: The size of the latent reservoir from each participant was measured by limiting dilution co-culture assay two weeks before and ten weeks after disulfiram administration..
Measure: Mean (95% Confidence Interval); unit: Fold change in IUPM
Units Other Than Participants: Blood samples
Arm/Group | Intervention Arm
Number analyzed (Participants) | 16
Number analyzed (Blood samples) | 32
Fold change in IUPM | 1.16 [0.70 to 1.92]

2. Primary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of a two-week course of disulfiram was defined using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). Details are available on the RSC website (http://rsc.tech-res.com/safetyandpharmacovigilance/). The number of adverse events and their grade was determined for each subject.
Time Frame: Two weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 16
Participants | 0

3. Primary Outcome: The Fold Change in Mean Levels of Viremia During and After Disulfiram Dosing as Compared to Baseline Levels
Description: Residual viremia was measured using a singe copy assay (SCA) in plasma samples obtained at enrollment, Days -14, -7, 0, 2, 4, 7, 9, 11, 14, 16, and 18, and at weeks 3, 4, 8 and 12. The level of residual viremia measured by SCA prior to disulfiram (Days 14, 17 and 0), during treatment (Days 1 to 14) and after dosing (Days 16 and 18) was modelled using negative binomial regression, and reported as the mean fold-change during and after disulfiram as compared to that during the baseline period.
Time Frame: Baseline to Day 18
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Intervention Arm
Number analyzed (Participants) | 16
Fold change | 1.5 [0.9 to 2.7]

4. Primary Outcome: Number of Participants With Detectable Plasma HIV RNA
Description: Plasma HIV RNA levels were measured weekly using a commercial assay. The number of participants who had a detectable viral load (> 50 copies RNA/mL) was determined.
Time Frame: Two weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 16
Participants | 1

ADVERSE EVENTS:
Arm/Group | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No